CLINICAL TRIAL: NCT00690170
Title: Nicotinic Modulation of (NMDA) Receptor Antagonist Schizophrenia-like Information Processing Deficits in Humans
Brief Title: Nicotinic Modulation of Schizophrenia-like Information Processing Deficits in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18014
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects
Keywords: ketamine; nicotine; schizophrenia; cognitive deficits; P300 oddball paradigm; Mismatch Negativity; P50 gating
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Ketamine; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ketamine and Nicotine (Active Comparator): * 0.23 mg/kg of ketamine bolus IV (in the arm) over one minute followed by maintenance infusion at 0.58mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 64 minutes.
  * 13.5 µg/kg of nicotine IV (in the arm) given over 10 min (1.35 µg/min/kg), followed by a constant infusion of 31.02 µg/kg given over 85 min (0.365 µg/min/kg)
  Interventions: Drug: Ketamine and Nicotine
- Placebo Comparator (Placebo Comparator): -Placebo administration: Normal saline (sodium chloride 0.9%)over 95 minutes
  Interventions: Drug: Placebo
- Ketamine and Placebo (Active Comparator): Ketamine administration: 0.23 mg/kg bolus over one minute followed by maintenance infusion at 0.58mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 64 minutes
  Placebo administration: Normal saline (sodium chloride 0.9%)over 94 minutes
  Interventions: Drug: Ketamine
- Nicotine and Placebo (Active Comparator): Nicotine: 13.5 µg/kg given over 10 min (1.35 µg/min/kg)IV (in the arm), followed by a constant infusion of 31.02 µg/kg given over 85 min (0.365 µg/min/kg) Placebo: Normal saline (sodium chloride 0.9%)IV (in the arm)
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Ketamine — Ketamine: 0.23 mg/kg bolus over one minute followed by maintenance infusion at 0.58mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 64 minutes
  Other Names: K; Special K
  Arms: Ketamine and Placebo
Drug: Nicotine — Nicotine: 13.5 µg/kg given over 10 min (1.35 µg/min/kg),IV (in the arm) followed by a constant infusion of 31.02 µg/kg given over 85 min (0.365 µg/min/kg) Placebo: Normal saline (sodium chloride 0.9%)IV (in the arm)
  Arms: Nicotine and Placebo
Drug: Placebo — Normal saline (sodium chloride 0.9%)administered via IV (in the arm) over 95 minutes
  Arms: Placebo Comparator
Drug: Ketamine and Nicotine — 0.23 mg/kg of ketamine bolus IV (in the arm) over one minute followed by maintenance infusion at 0.58mg/kg/hour x 30 minutes, followed by 0.29 mg/kg/hour x 64 minutes.
  13.5 µg/kg of nicotineIV (in the arm) given over 10 min (1.35 µg/min/kg), followed by a constant infusion of 31.02 µg/kg given over 85 min (0.365 µg/min/kg)
  Arms: Ketamine and Nicotine

SUMMARY:
This study examines the interactive effects of ketamine and nicotine.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2002-12; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
ERP recording procedures: Brain wave activity during tasks involving in processing auditory and visual stimuli with different degrees of attentional and memory demands will be recorded. | +65
IntegNeuro is a computerized battery that consists of an automated stimulus presentation to measure cognitive function. | +25
Positive and Negative Syndrome Scale will be used to measure psychotic symptoms. | -90, +10, +105, +180

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Veterans Administration Hospital, West Haven, Connecticut, United States

REFERENCES:
- [Derived] D'Souza DC, Ahn K, Bhakta S, Elander J, Singh N, Nadim H, Jatlow P, Suckow RF, Pittman B, Ranganathan M. Nicotine fails to attenuate ketamine-induced cognitive deficits and negative and positive symptoms in humans: implications for schizophrenia. Biol Psychiatry. 2012 Nov 1;72(9):785-94. doi: 10.1016/j.biopsych.2012.05.009. Epub 2012 Jun 19. PMID 22717030